CLINICAL TRIAL: NCT03471416
Title: Nutritional Status in Children With Acute Lymphoblastic Leukemia (ALL) Undergoing Treatment at the National Pediatric Oncology Unit in Guatemala City, Guatemala
Brief Title: Nutritional Status in Children With ALL in Guatemala
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Unidad nacional de Oncologia Pediatrica, Guatemala (Other)
Responsible Party: Sponsor
Other Study IDs: AAAR4744
Record Dates: First submitted 2018-03-14; First posted 2018-03-20 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Guatemala; Guatemala City; Malnutrition; Leukemia; Childhood Cancer
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Malnutrition; Leukemia; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with ALL: Children undergoing ALL treatment at UNOP Guatemala who are under the age of 18 years.
- Healthy siblings: Healthy siblings of children undergoing ALL treatment at UNOP Guatemala who are under the age of 18 years.

SUMMARY:
This study proposes to investigate the association of nutritional status of a children assessed by body mass index (BMI), triceps skinfold thickness (TSFT), and mid upper arm circumference (MUAC), with body composition, measured by dual-energy X-ray absorptiometry (DEXA), in 60 children undergoing treatment of ALL at Unidad Nacional de Oncologia Pediatrica (UNOP), in Guatemala City, Guatemala. The study also aims to establish normative values of body composition in children residing in an LMIC by examining 160 healthy siblings of children under treatment, and to measure habitual physical activity in children with acute lymphoblastic leukemia (ALL) at diagnosis and during therapy.

DETAILED DESCRIPTION:
The majority of children with cancer live in low and middle income countries (LMICs) where malnutrition, both under and over nutrition, is highly prevalent. Children who are malnourished while undergoing treatment for acute lymphoblastic leukemia (ALL) are shown to have chances of reduced survival. Children, who are malnourished at diagnosis, if the nutritional status is improved over the course of 6 months during the ALL treatment, have chances of similar survival as the ones who were nourished throughout. Therefore, it is important to study nutritional status in children with ALL, to understand and implement better treatment outcomes. Height and weight alone are considered incomprehensive in classifying nutritional status, especially in poorly nourished children. A more advanced nutritional assessment that distinguishes between fat and muscle mass is required. Treatment for ALL results in an increase in weight over the course of therapy with preferential gain in fat mass (FM) compared to fat free mass (FFM). Hence, there is a pressing need to advance nutritional assessment and implementation in pediatric oncology that includes monitoring of FM and FFM.

ELIGIBILITY:
Inclusion Criteria:

* Children under treatment for Acute Lymphoblastic Leukemia (ALL)
* Age under 18 years
* Getting treatment at UNOP

Exclusion Criteria:

* If they can't participate in the study due to illness or long distance to travel to UNOP

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children undergoing ALL treatment at UNOP Guatemala - must be under the age of 18 years. Their healthy siblings will be recruited to compare body composition.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Association of BMI and Body Composition | Up to 6 months after treatment
  Body composition will be measured by DEXA.
Association of TSFT and Body Composition | Up to 6 months after treatment
  Body composition will be measured by DEXA.
Association of MUAC and Body Composition | Up to 6 months after treatment
  Body composition will be measured by DEXA.

SECONDARY OUTCOMES:
Body Composition | Up to 6 months after treatment
  Aim to establish normative values of body composition (measured by DEXA) in children residing in an LMIC by examine healthy siblings of children under treatment at UNOP.
Habitual Activity Estimation Scale | Up to 6 months after treatment
  Percentage of time awake will be documented in each of 4 activity categories: inactive (lying down), somewhat inactive (SI, sitting down), somewhat active (SA, walking) and very active (VA, those activities that make subject "breathe hard and sweat"). The use of wake-up and bedtimes as well as meal times and durations allow the calculation of the total number of hours per day spent in each of the 4 categories. Total activity (TA) is calculated as SA+VA for each day.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Barr, MB, ChB, MD, Study Chair — McMaster University; Federico Antiloon, MD, MMM, PhD, Principal Investigator — Unidad Nacional de Oncología Pediátrica; Elena J Ladas, RD, PhD, Study Director — Columbia University
Locations (1):
- Unidad Nacional de Oncología Pediátrica (UNOP), Guatemala City, Guatemala

IPD SHARING:
Plan to Share IPD: Undecided
The database is secured in Guatemala research site at UNOP. De-identified data is shared with Columbia University Medical Center via REDCap database system - managed by Columbia University.